CLINICAL TRIAL: NCT04836481
Title: A Pharmacokinetic Analysis of Levetiracetam Prophylaxis in Critically Ill Patients With Severe Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: American College of Clinical Pharmacy (Other)
Responsible Party: Principal Investigator, Sarah Schuman Harlan, Pharmacy Resident, Primary Investigator, University of Cincinnati
Other Study IDs: 2020-0744
Record Dates: First submitted 2020-12-10; First posted 2021-04-08 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injury
Keywords: Levetiracetam; Seizure Prophylaxis; Pharmacokinetic
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- LEV8: Levetiracetam 1000 mg every 8 hours
  Interventions: Other: Serum Sample Collection
- LEV12: Levetiracetam 1000 mg every 12 hours
  Interventions: Other: Serum Sample Collection

INTERVENTIONS:
Other: Serum Sample Collection — Each patient will have 5 serum samples collected for analysis after a minimum six consecutive doses. Patients receiving LEV8 will have sampled collected at hours 0.5, 1, 4, 6, and 8. Patients receiving LEV12 will have sampled collected at hours 0.5, 1, 4, 8, and 12.

SUMMARY:
This study aims is to describe the pharmacokinetic properties of levetiracetam through measurement of serum concentrations in critically ill, severe traumatic brain injury patients.

DETAILED DESCRIPTION:
Levetiracetam (LEV) is widely used for the prevention and treatment of seizures given its favorable pharmacokinetic profile. A strong correlation between serum concentrations and clinical efficacy has yet to be established; however, a target of 6-20 g/mL is recommended. Limited evidence exists supporting an optimal dosing strategy to achieve these target concentrations in neurocritically ill patients. Previous pharmacokinetic models suggest LEV 1000 mg every 8 hours achieves the highest proportion of therapeutic serum concentrations, but this dosing strategy has not been clinically studied in neurocritically ill patients. Additionally, only one phase two study has evaluated LEV pharmacokinetics in severe traumatic brain injury (TBI).

The aim of this study is to describe the pharmacokinetic properties of LEV through measurement of serum concentrations in critically ill, severe TBI patients. Secondarily, this study aims to develop a population pharmacokinetic model aimed at characterizing LEV dose optimization in severe TBI. An exploratory aim is to evaluate LEV pharmacodynamics in severe TBI patients through evaluation of physiologic, electrophysiologic and biochemical changes using multimodal monitoring or surface electroencephalogram (EEG), as available. A subgroup analysis will evaluate LEV pharmacokinetics in severe TBI patients with augmented renal clearance (ARC).

This prospective, single-center pharmacokinetic and pharmacodynamic study will include critically ill patients receiving intravenous LEV for seizure prophylaxis following severe TBI. Patients with severe TBI qualifying for multimodal monitoring will receive LEV 1000 mg every 8 hours (LEV8) per institutional practice. All other severe TBI patients will receive LEV 1000 mg every 12 hours (LEV12) according to institution practice. Patients with renal dysfunction (creatinine clearance < 50 mL/min) will be excluded. All patients will have five serum samples collected following the sixth or greater consecutive dose. Patients receiving LEV8 will have samples collected at 0.5, 1, 4, 6, and 8 hours. Patients receiving LEV12 will have samples collected at 0.5, 1, 4, 8, and 12 hours. Serum concentrations will be analyzed with pharmacokinetic modeling and Monte Carlo simulations. LEV pharmacodynamics will be evaluated in patients receiving multimodal monitoring or surface EEG, as available. Analysis of ARC will include patients with Augmented Renal Clearance in Trauma Intensive Care (ARTIC) score >6 during sampling.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the neurosurgical intensive care unit or surgical intensive care unit following severe traumatic brain injury (post-resuscitation GCS 3-8 with or without CT abnormalities)
* Receiving intravenous levetiracetam for seizure prophylaxis at a dose of 1000 mg every 12 hours or 1000 mg every 8 hours at time of enrollment

Exclusion Criteria:

* Known history of epilepsy or seizure disorder
* Taking antiseizure medication prior to admission
* Taking medication with known effect on levetiracetam pharmacokinetics including carbamazepine, phenytoin, oxcarbazepine, mefloquine, methotrexate, mianserin, or orlistat
* Weight < 50 kg
* Anticipated survival <72 hours from injury, as deemed by the primary neurosurgical provider
* Acute Kidney Injury (Scr rise > 0.3 mg/dL from baseline) or creatinine clearance <50 mL/min at time of enrollment
* Prisoners
* Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study will be patients with severe traumatic brain injury, defined as a post-resuscitation GCS 3-8 with or without CT abnormalities who are receiving intravenous levetiracetam 1000 mg every 8 or every 12 hours for seizure prophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Serum Levetiracetam Concentration 1 | Hour 0.5
  Serum levetiracetam concentration collected at 0.5 hours after target dose for sampling
Serum Levetiracetam Concentration 2 | Hour 1
  Serum levetiracetam concentration collected at hour 1 after target dose for sampling
Serum Levetiracetam Concentration 3 | Hour 4
  Serum levetiracetam concentration collected at hour 4 after target dose for sampling
Serum Levetiracetam Concentration 4 | Hour 6-8
  Serum levetiracetam concentration collected at hour 6 (patients receiving every 8 hour levetiracetam) or hour 8 (patients receiving every 12 hour levetiracetam)
Serum Levetiracetam Concentration 5 | Hour 8-12
  Serum levetiracetam concentration collected at hour 8 (patients receiving every 8 hour levetiracetam) or hour 12 (patients receiving every 12 hour levetiracetam)

SECONDARY OUTCOMES:
Intracranial Pressure | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
Cerebral Perfusion Pressure | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
Pressure Reactivity Index | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
Cerebral Blood Flow | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
Cerebral Microdialysis Glucose Concentration | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
Cerebral Microdialysis Pyruvate Concentration | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
Cerebral Microdialysis Lactate Concentration | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
Cerebral Microdialysis Glutamate Concentration | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
Cerebral Microdialysis Glycerol Concentration | Baseline to Day 7
  Collected at baseline and at each time of serum sample collection for pharmacodynamic analysis
ARTIC Score | Hour 0.5 (Collected at time of first serum sample collection)
  Calculated ARTIC score

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Schuman Harlan, PharmD, Principal Investigator — University of Cincinnati; Shaun Keegan, PharmD, Principal Investigator — University of Cincinnati; Carolyn Philpott, PharmD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cook AM, Hatton-Kolpek J. Augmented Renal Clearance. Pharmacotherapy. 2019 Mar;39(3):346-354. doi: 10.1002/phar.2231. Epub 2019 Mar 11. PMID 30723936
- [Background] Rowe AS, Goodwin H, Brophy GM, Bushwitz J, Castle A, Deen D, Johnson D, Lesch C, Liang N, Potter E, Roels C, Samaan K, Rhoney DH; Neurocritical Care Society Pharmacy Section. Seizure prophylaxis in neurocritical care: a review of evidence-based support. Pharmacotherapy. 2014;34(4):396-409. doi: 10.1002/phar.1374. Epub 2013 Nov 26. PMID 24277723
- [Background] Barletta JF, Mangram AJ, Byrne M, Sucher JF, Hollingworth AK, Ali-Osman FR, Shirah GR, Haley M, Dzandu JK. Identifying augmented renal clearance in trauma patients: Validation of the Augmented Renal Clearance in Trauma Intensive Care scoring system. J Trauma Acute Care Surg. 2017 Apr;82(4):665-671. doi: 10.1097/TA.0000000000001387. PMID 28129261
- [Result] Zangbar B, Khalil M, Gruessner A, Joseph B, Friese R, Kulvatunyou N, Wynne J, Latifi R, Rhee P, O'Keeffe T. Levetiracetam Prophylaxis for Post-traumatic Brain Injury Seizures is Ineffective: A Propensity Score Analysis. World J Surg. 2016 Nov;40(11):2667-2672. doi: 10.1007/s00268-016-3606-y. PMID 27307089
- [Result] Gabriel WM, Rowe AS. Long-term comparison of GOS-E scores in patients treated with phenytoin or levetiracetam for posttraumatic seizure prophylaxis after traumatic brain injury. Ann Pharmacother. 2014 Nov;48(11):1440-4. doi: 10.1177/1060028014549013. Epub 2014 Aug 28. PMID 25169249
- [Result] Inaba K, Menaker J, Branco BC, Gooch J, Okoye OT, Herrold J, Scalea TM, Dubose J, Demetriades D. A prospective multicenter comparison of levetiracetam versus phenytoin for early posttraumatic seizure prophylaxis. J Trauma Acute Care Surg. 2013 Mar;74(3):766-71; discussion 771-3. doi: 10.1097/TA.0b013e3182826e84. PMID 23425733
- [Result] Jones KE, Puccio AM, Harshman KJ, Falcione B, Benedict N, Jankowitz BT, Stippler M, Fischer M, Sauber-Schatz EK, Fabio A, Darby JM, Okonkwo DO. Levetiracetam versus phenytoin for seizure prophylaxis in severe traumatic brain injury. Neurosurg Focus. 2008 Oct;25(4):E3. doi: 10.3171/FOC.2008.25.10.E3. PMID 18828701
- [Result] Szaflarski JP, Sangha KS, Lindsell CJ, Shutter LA. Prospective, randomized, single-blinded comparative trial of intravenous levetiracetam versus phenytoin for seizure prophylaxis. Neurocrit Care. 2010 Apr;12(2):165-72. doi: 10.1007/s12028-009-9304-y. PMID 19898966
- [Result] Ramael S, Daoust A, Otoul C, Toublanc N, Troenaru M, Lu ZS, Stockis A. Levetiracetam intravenous infusion: a randomized, placebo-controlled safety and pharmacokinetic study. Epilepsia. 2006 Jul;47(7):1128-35. doi: 10.1111/j.1528-1167.2006.00586.x. PMID 16886975
- [Result] Steinhoff BJ, Staack AM. Levetiracetam and brivaracetam: a review of evidence from clinical trials and clinical experience. Ther Adv Neurol Disord. 2019 Sep 9;12:1756286419873518. doi: 10.1177/1756286419873518. eCollection 2019. PMID 31523280
- [Result] Spencer DD, Jacobi J, Juenke JM, Fleck JD, Kays MB. Steady-state pharmacokinetics of intravenous levetiracetam in neurocritical care patients. Pharmacotherapy. 2011 Oct;31(10):934-41. doi: 10.1592/phco.31.10.934. PMID 21950640
- [Result] Cotta MO, Abdul-Aziz MH, Frey OR, Sime FB, Roberts JA, Roehr AC. What Are the Predictors for Achieving Therapeutic Levetiracetam Serum Concentrations in Adult Neurological Patients? Ther Drug Monit. 2020 Aug;42(4):626-630. doi: 10.1097/FTD.0000000000000731. PMID 31977751
- [Result] Klein P, Herr D, Pearl PL, Natale J, Levine Z, Nogay C, Sandoval F, Trzcinsky S, Atabaki SM, Tsuchida T, van den Anker J, Soldin SJ, He J, McCarter R. Results of phase II pharmacokinetic study of levetiracetam for prevention of post-traumatic epilepsy. Epilepsy Behav. 2012 Aug;24(4):457-61. doi: 10.1016/j.yebeh.2012.05.011. Epub 2012 Jul 7. PMID 22771222
- [Result] Uges JW, van Huizen MD, Engelsman J, Wilms EB, Touw DJ, Peeters E, Vecht CJ. Safety and pharmacokinetics of intravenous levetiracetam infusion as add-on in status epilepticus. Epilepsia. 2009 Mar;50(3):415-21. doi: 10.1111/j.1528-1167.2008.01889.x. Epub 2008 Nov 17. PMID 19054418
- [Result] Udy A, Boots R, Senthuran S, Stuart J, Deans R, Lassig-Smith M, Lipman J. Augmented creatinine clearance in traumatic brain injury. Anesth Analg. 2010 Dec;111(6):1505-10. doi: 10.1213/ANE.0b013e3181f7107d. Epub 2010 Nov 3. PMID 21048095
- [Result] May CC, Arora S, Parli SE, Fraser JF, Bastin MT, Cook AM. Augmented Renal Clearance in Patients with Subarachnoid Hemorrhage. Neurocrit Care. 2015 Dec;23(3):374-9. doi: 10.1007/s12028-015-0127-8. PMID 25761425
- [Result] Tong X, Patsalos PN. A microdialysis study of the novel antiepileptic drug levetiracetam: extracellular pharmacokinetics and effect on taurine in rat brain. Br J Pharmacol. 2001 Jul;133(6):867-74. doi: 10.1038/sj.bjp.0704141. PMID 11454660
- [Result] Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron. 1976;16(1):31-41. doi: 10.1159/000180580. PMID 1244564